CLINICAL TRIAL: NCT00425464
Title: A Prospective Multicenter Clinical Study to Evaluate the Safety and Effectiveness of the Synchrony Dual Optic Intraocular Lens in Patients Undergoing Cataract Extraction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYNC-601-IOL
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

ARMS (2):
- Synchrony® Dual Optic Intraocular Lens (Experimental)
  Interventions: Device: Synchrony® Dual Optic Intraocular Lens
- Standard Monofocal Intraocular Lens (Active Comparator)
  Interventions: Device: Standard Monofocal Intraocular Lens

INTERVENTIONS:
Device: Standard Monofocal Intraocular Lens — The control (active comparator) arm is comprised of patients who meet all study eligibility criteria and will be implanted with a standard monofocal intraocular lens.
  Each study patient will undergo standard extracapsular cataract extraction through a clear corneal or limbal incision and circular continuous curvilinear capsulorhexis.
  Arms: Standard Monofocal Intraocular Lens
Device: Synchrony® Dual Optic Intraocular Lens — The Synchrony® Dual Optic Intraocular Lens (experimantal) arm is comprised of patients who meet all study eligibility criteria and will be implanted with a Synchrony® Dual Optic Intraocular Lens.
  Each study patient will undergo standard extracapsular cataract extraction through a clear corneal or limbal incision and circular continuous curvilinear capsulorhexis.
  Arms: Synchrony® Dual Optic Intraocular Lens

SUMMARY:
The purpose of the study is to determine if the Synchrony Dual Optic Accommodating Intraocular Lens can be used safely and effectively in post cataract extraction subjects

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be scheduled to undergo primary intraocular lens implantation for the correction of aphakia following extraction of a senile cataract.
2. Patients must have a cataract causing reduction in visual acuity to a level of 20/40 or worse with BAT on medium setting.
3. Patients must require Synchrony® Lens correction of 16D - 28D or, if participating in the control study, patients must require a Clariflex® (AMO®), Phacoflex® II models SI30NB (AMO®) or a SI40NB (AMO®).
4. Patients must have ≤ 1.0 D of preoperative keratometric astigmatism.
5. Patients must have clear intraocular media other than cataract(s).
6. Patients must be age 50 or older at the time of implantation.
7. Patient must be willing and able to return for all scheduled follow-up examinations and have signed a written informed consent form.

Exclusion Criteria:

1. Patients with any anterior segment pathology (anterior segment or corneal abnormalities, chronic uveitis, iritis, corneal dystrophy, pseudoexfoliation, etc.).
2. Patients with glaucoma, glaucoma suspect or ocular hypertension, i.e., IOP > 22 mmHg.
3. Patients with previous retinal detachment or retinal pathology including age- related macular degeneration.
4. Patients with diabetes, currently being treated systemically.
5. Patients with systemic or ocular disease that may prevent the patient from achieving uncorrected distance visual acuity of 20/32 or better post operatively.
6. Patients with congenital bilateral cataract.
7. Patients who require chronic administration of any topical ophthalmic or systemic medication that may affect accommodation such as mydriatic, cycloplegic and myotic agents; tricyclic antidepressants, phenothiazines, benzodiazepines, first generation antihistamines, anticholinergic agents. The use of tamsulosin hydrochloride (Flomax®) is also excluded preoperatively due to floppy iris syndrome.
8. Patients with best corrected visual acuity of 20/80 or worse in the fellow eye not attributable to cataract.
9. Patients who are currently participating or have participated in an investigational study, other than this study, within the past 60 days.
10. Patients who have had previous ocular surgery in the operative eye, including refractive surgery.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2005-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Distance corrected near visual acuity | 1 Mo, 4-6 Mo, 12 Mo, 24 Mo, & 36 Mo

SECONDARY OUTCOMES:
Best corrected distance visual acuity | 1 Mo, 4-6 Mo, 12 Mo, 24 Mo, & 36 Mo

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Harvard Eye Associates, Laguna Hills, California
  - Long Beach Laser Center, Los Alamitos, California
  - Altos Eye Physicians, Los Altos, California
  - Grutzmacher & Lewis, Sacramento, California
  - Davidorf Eye Group, West Hills, California
  - Glaucoma Consultants of Colorado, Parker, Colorado
  - Katzen Eye Care and Laser Center, Boynton Beach, Florida
  - EyeSight Hawaii, Honolulu, Hawaii
  - The Midwest Center for Sight, Des Plaines, Illinois
  - NorthShore University HealthSystem, Glenview, Illinois
  - Wallace Eye Surgery, Alexandria, Louisiana
  - Chu Vision Institute, Bloomington, Minnesota
  - Associated Eye Care, Stillwater, Minnesota
  - Pepose Vision Institute, Chesterfield, Missouri
  - Nevada Eye Care, Las Vegas, Nevada
  - Drs. Fine, Hoffman & Packer, Eugene, Oregon
  - Alkek Eye Center, Houston, Texas
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - Northwest Eye Surgeons, Seattle, Washington
  - Davis Duehr Dean, Madison, Wisconsin